CLINICAL TRIAL: NCT06221657
Title: A Single-center, Prospective, Randomized, Open-label, Comparative, Investigator-initiated Clinical Trial to Confirm the Non-inferiority and Safety of Tenofovir Alafenamide and Tenofovir Disoproxil Fumarate in Patients With Hematologic Malignancies Who Require Prophylactic Hepatitis B Antiviral Treatment
Brief Title: Clinical Trial for Non-inferiority and Safety of Tenofovir Alafenamide and Tenofovir Disoproxil Fumarate in Patients With Hematologic Malignancies Who Require Prophylactic Hepatitis B Antiviral Treatment
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Hye Won Lee, professor, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IIT-TAF-01
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Patients With Malignant Blood Disease Requiring Hepatitis B Antiviral Medication
MeSH Terms: interventions — tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAF group (Experimental)
  Interventions: Drug: Vemlidy
- TDF group (Active Comparator)
  Interventions: Drug: Virreal

INTERVENTIONS:
Drug: Vemlidy — 1 tablet once a day, oral administration
  Arms: TAF group
Drug: Virreal — 1 tablet once a day, oral administration
  Arms: TDF group

SUMMARY:
his clinical trial was conducted to determine the non-inferiority and safety of prophylactic antiviral treatment of Tenofovir alafenamide (TAF) compared to Tenofovir disoproxil fumarate (TDF) in patients with malignant hematological diseases requiring prophylactic hepatitis B antiviral treatment. Confirm.

In the case of TAF, domestic evidence when used as a first-line treatment is insufficient, so in this clinical trial, the virus suppression effect compared to TDF during the first administration of TAF to patients with malignant hematological diseases requiring prophylactic hepatitis B antiviral treatment was investigated. We aim to secure non-inferiority and additionally confirm the safety of TAF's known advantages of reducing renal function damage and protecting bone function.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women over 19 years of age and under 65 years of age
2. Patients who meet the following criteria A or B A. Those scheduled for hematopoietic stem cell transplantation and treatment with immunosuppressants or chemotherapy.

   B. Those scheduled to receive anticancer treatment including rituximab
3. HBcAb positive patient
4. Patients who voluntarily agreed to participate in this clinical trial and signed a written consent form

Exclusion Criteria:

1. Patients taking oral chronic hepatitis B antiviral drugs before starting the study
2. Galactose intolerance. Patients with genetic problems such as Lapp lactase deficiency or glucose-galactose malabsorption
3. Patients with hypersensitivity to tenofovir alafenamide citrate or tenofovir disoproxil orotate
4. Patients with abnormal renal function (e-GFR less than 15mL/min) or end-stage renal disease requiring dialysis
5. Hepatitis C patients
6. HIV-infected patients
7. Pregnant women, lactating women, or patients planning to become pregnant
8. If you are participating in another clinical trial administering medication
9. Patients who do not agree to participate in this clinical trial
10. Adults with impaired consent capacity who are unable to give consent on their own
11. Those who have taken other clinical trial drugs for less than 24 weeks
12. Other clinically determined by the principal investigator to be difficult for the clinical trial subject to conduct the clinical trial.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects maintained at HBV DNA <29 IU/mL | 48 weeks

SECONDARY OUTCOMES:
Proportion of subjects maintaining HBV DNA <29 IU/mL | 72 weeks
Proportion of subjects with serum HBV DNA <60 IU/mL | 12, 24, 48, 72 weeks
Proportion of subjects maintaining HBV DNA <10 IU/mL | 12, 24, 48, 72 weeks
Level of AST, ALT, r-GTP | 12, 24, 48, 72 weeks
total cholesterol, LDL-cholesterol, HDL-cholesterol, triglyceride | 12, 24, 48, 72 weeks
level of e-GFR | 12, 24, 48, 72 weeks
creatinine clearance rate | 12, 24, 48, 72 weeks
BMD T Score | 24, 48, 72 weeks
blood Phosphorus levels | 12, 24, 48, 72 weeks

IPD SHARING:
Plan to Share IPD: No